CLINICAL TRIAL: NCT00204048
Title: A Multicenter Trial of Academic Hospitalists
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 9967
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: Hospitalists
MeSH Terms: interventions — Behavior Observation Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Observation (behavior) — Inpatients admitted in GenMed at the University of Chicago will be consented to participate in an inpatient interview that consists of questions related to quality of care and satisfaction. The patient will also be interviewed over the phone 30 days after discharge and will be asked questions related to current health and their satisfaction during their stay at University of Chicago.

SUMMARY:
Care of hospitalized patients by "hospitalists" -- often defined as physicians who dedicate at least 25% of their practice to inpatient care -- is a recent, growing, and controversial trend in health care delivery in the United States. But despite the growth of interest in hospitalists, there have been few scientific evaluations of the concept. The comprehensive aim of this research study is to measure and analyze the effects of hospitalists on patient outcomes, costs and medical education on the general medical services of a group of academic centers.

DETAILED DESCRIPTION:
In 2001, a study titled, "A Multi-Center Trial of Academic Hospitalists" began at the University of Chicago Hospital along with five additional academic institutions. The study is currently and successfully collecting data solely at the University of Chicago Medical Center.

The comprehensive aim of this proposed research is to measure and analyze the effects of hospitalists on patient outcomes, costs, and medical education on the general medicine services at the University of Chicago Medical Center (UC). The comprehensive aim of this research will be pursued through five specific aims:

Specific Aim #1- To assess whether hospitalists affect the cost and quality of inpatient care. This will be accomplished by analyzing the outcomes of 50,000 patients assigned to hospitalists or non-hospitalists using a quasi-randomized design based on day of the week of admission. Outcomes will include in-hospital and post-discharge mortality, readmission, emergency room use, and patient satisfaction.

Specific Aim #2- To assess the mechanisms by which hospitalists may effect the cost and quality of care. Understanding these mechanisms is essential if hospitalist programs are to be designed in ways that permit them to achieve their desired benefits. We will develop measures to assess the whether these possible mechanisms by which hospitalists may have their effects are related to costs and outcomes.

Specific Aim #3- To assess the effects of hospitalists on housestaff and student education and satisfaction. This will be accomplished by surveys administered to medical students and housestaff.

Specific Aim #4 - To attempt to quantify primary care providers' (PCP's) satisfaction with the frequency, promptness, manner, and content of communication with the in-hospital healthcare team, and to assess differences in PCP satisfaction with teams led by hospitalist and non-hospitalist attending physicians. We hypothesize that deficiencies in such communication may impair continuity of care with outpatient physicians during hospitalization and at the time of discharge, and may be improved when the attending physician is a hospitalist.

Specific Aim #5- To assess the quality of care for vulnerable elders for specific geriatric syndromes and diseases by modifying our current surveys and chart abstraction tools in our project with questions aimed to address these issues.

ELIGIBILITY:
Inclusion Criteria:

* General Medicine inpatients at the University of Chicago Hospital or Mercy Hospital in Chicago Illinois

Exclusion Criteria:

* Non-General Medicine inpatients

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients admitted in General Medicine at the University of Chicago
Sampling Method: Probability Sample
Enrollment: 104940 (Actual)
Dates: Start 2001-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
the effects of hospitalists on patient outcomes, costs, and medical education on the general medicine services | 30 days after discharge
  This will be accomplished by analyzing the outcomes of 60,000 patients assigned to hospitalists or non-hospitalists using a quasi-randomized design based on day of the week of admission. Outcomes will include in-hospital and post-discharge mortality, readmission, emergency room use, and patient satisfaction

SECONDARY OUTCOMES:
the effects of hospitalists on housestaff and student education and satisfaction | 1 academic year
  This will be accomplished by surveys administered to medical students and housestaff.
quality of care for vulnerable elders | 30 days after discharge
  chart abstraction tools in our project with questions aimed to address these issues

CONTACTS AND LOCATIONS:
Overall Officials: David Meltzer, M.D., Ph.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karliner LS, Kim SE, Meltzer DO, Auerbach AD. Influence of language barriers on outcomes of hospital care for general medicine inpatients. J Hosp Med. 2010 May-Jun;5(5):276-82. doi: 10.1002/jhm.658. PMID 20533573
- [Derived] Hasan O, Meltzer DO, Shaykevich SA, Bell CM, Kaboli PJ, Auerbach AD, Wetterneck TB, Arora VM, Zhang J, Schnipper JL. Hospital readmission in general medicine patients: a prediction model. J Gen Intern Med. 2010 Mar;25(3):211-9. doi: 10.1007/s11606-009-1196-1. Epub 2009 Dec 15. PMID 20013068
- [Derived] Auerbach AD, Katz R, Pantilat SZ, Bernacki R, Schnipper J, Kaboli P, Wetterneck T, Gonzales D, Arora V, Zhang J, Meltzer D. Factors associated with discussion of care plans and code status at the time of hospital admission: results from the Multicenter Hospitalist Study. J Hosp Med. 2008 Nov-Dec;3(6):437-45. doi: 10.1002/jhm.369. PMID 19084893
- [Derived] Vasilevskis EE, Meltzer D, Schnipper J, Kaboli P, Wetterneck T, Gonzales D, Arora V, Zhang J, Auerbach AD. Quality of care for decompensated heart failure: comparable performance between academic hospitalists and non-hospitalists. J Gen Intern Med. 2008 Sep;23(9):1399-406. doi: 10.1007/s11606-008-0680-3. Epub 2008 Jul 1. PMID 18592321